CLINICAL TRIAL: NCT00102570
Title: Clinical and Immunological Evaluation of Children With Allergic Disease
Brief Title: Clinical and Immunological Evaluation of Children With Allergies
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 050084; 05-I-0084
Record Dates: First submitted 2005-01-29; First posted 2005-01-31 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2010-08-10

CONDITIONS: Hypersensitivity, Immediate
Keywords: Pediatric; Atopic; Asthma; Rhinitis; Outpatient; Allergy; Pediatric Allergy; Food Allergy; Stinging Insect Allergy; Atopic Dermatitis; Insect Sting
MeSH Terms: conditions — Hypersensitivity, Immediate; Asthma; Rhinitis; Hypersensitivity; Food Hypersensitivity; Dermatitis, Atopic; Insect Bites and Stings

SUMMARY:
This study will evaluate children with allergies and collect medical data and biological specimens from them periodically to learn more about the diseases and gain information that may be useful in developing new treatments.

Patients 6 months to 18 years of age with a possible diagnosis of asthma, rhinitis, anaphylaxis, hives, atopic dermatitis, food allergy, stinging insect allergy, and other allergic and inflammatory diseases may be eligible for this study. Biological parents of patients may also be enrolled to provide a blood sample for genetic studies.

Participants undergo tests appropriate for the diagnosis and management of their allergy. They include the tests outlined below and, when necessary, additional blood tests, tissue biopsies (surgical removal of a small piece of tissue for microscopic examination), computed tomography (CT) or magnetic resonance imaging (MRI).

* Pulmonary function test: This test evaluates lung function. The patient blows hard into a tube attached to a machine to measure the airflow from the lungs. At home, the patient uses a small plastic device called a peak flow meter to measure lung function. Patients whose lung function measures less than 80 percent the value predicted for his or her age may be given the medicine albuterol to see if lung function improves.
* Skin prick testing: Drops of up to 55 different allergens (foreign substances, such as pollen and certain foods or medicines that cause reactions like sneezing, hives, eczema, and others) are placed on the back or arm. The skin under the allergen is then scratched with a pointed tool. If the person is allergic, the skin around the scratch develops a small area of itching, redness, or swelling that goes away after 30 to 60 minutes.
* Acoustic rhinometry: To learn the effect of allergies on the size of the nasal cavity, the nasal canal size is measured by placing a small round probe on the nostril. The device sends out and receives a sound wave signal from which the size of the nasal canal is calculated, recorded and stored graphically on a computer screen. The procedure is repeated three times with each nostril.
* Computerized assessment of learning and mood: Patients who are age 10 or older may take this computer test to find out if allergies affect learning and mood. The test measures the child's ability to understand directions, solve problems, and remember things. It also includes questions about how the child feels in general.
* Behavioral assessment system for children: Patients who are age 8 or older may take this true/false questionnaire to assess mood.
* Blood may be drawn for the following purposes: in lieu of skin prick testing to determine sensitivity to allergens; to look for reasons for the severity or cause of an allergy; for research studies on the immune system, including markers of allergy; for genetic tests to determine inherited factors that increase the risk of developing allergies.

Patients are scheduled for follow-up visits based on their diagnosis and severity of illness. Most patients return for within one month of their first study visit and then, in general, once a month when allergies are severe, and every few months when they are more stable. Visits include an updated history and physical examination, blood tests, and possibly some of the tests described above. Patients may also have intradermal skin testing, in which allergens that are used for skin prick testing are injected into the forearms or upper arms just below the surface of the skin.

Patients who test positive to allergens may be offered standard treatment with allergy shots.

DETAILED DESCRIPTION:
Atopic disorders, including but not limited to asthma, rhinitis, anaphylaxis, urticaria, atopic dermatitis, food allergy, and stinging insect allergy are exceedingly common in the pediatric population. The impact that these disorders have on health, educational and social activities and costs of medical care are profound and widespread. In order to understand disease and improve therapy, the study of pediatric allergy is justifiably an important health priority and the goal of this protocol. This purpose will be fostered through the following objectives: 1) To gather a database of clinical and immunological data and to better clinically and immunologically characterize disease onset, progression and remittance of these disorders; 2) to foster collaborative studies in pediatric allergic disease with other institutions and 3) to provide a cohort of pediatric patients for residents in the NIH Clinical Center/NIAID Allergy and Immunology training program. Up to 500 new patients will be enrolled to attain these goals. Patients will undergo screening history, physical examination, and clinical laboratory evaluation according to the standard of practice in the community. Although imaging studies and tissue biopsies will be performed only when clinically indicated, blood samples for cellular and biochemical studies may be collected for research purposes. Treatment plans will be individualized for each patient and the number and length of additional visits and diagnostic evaluations will vary accordingly. Standard immunotherapy for allergic disease may be offered. Through the assessment, analysis, and treatment of a large cohort of patients, we will better understand disease manifestations, trends, outcomes, and mechanisms of pediatric allergy and lay the groundwork for discovery of new therapeutic modalities.

ELIGIBILITY:
* INCLUSION CRITERIA:

Males and females, age 3 months to 19 years old, (less than 18 years old).

Individuals referred to the NIH with a diagnosis of asthma, rhinitis, anaphylaxis, urticaria, atopic dermatitis, food allergy, stinging insect allergy or other allergic/inflammatory diseases.

Subjects must maintain a primary physician for protocol related and non-related long-term follow-up and for any emergency medical treatment required.

INCLUSION CRITERIA FOR PARENTS:

Must be biological Parent

Must have a child with a diagnosis of allergic disease

EXCLUSION CRITERIA:

Inability to provide informed consent or assent. In the case of minors, unavailability of a parent or guardian.

EXCLUSION CRITERIA FOR PARENTS:

Non-biological parent

Ages: 3 Months to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 270 (Actual)
Dates: Start 2005-01-26; Study Completion 2010-08-10

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Stone KD. Atopic diseases of childhood. Curr Opin Pediatr. 2003 Oct;15(5):495-511. doi: 10.1097/00008480-200310000-00009. PMID 14508299
- [Background] Juniper EF. Quality of life in adults and children with asthma and rhinitis. Allergy. 1997 Oct;52(10):971-7. doi: 10.1111/j.1398-9995.1997.tb02416.x. PMID 9360747
- [Background] Weinmann S, Kamtsiuris P, Henke KD, Wickman M, Jenner A, Wahn U. The costs of atopy and asthma in children: assessment of direct costs and their determinants in a birth cohort. Pediatr Allergy Immunol. 2003 Feb;14(1):18-26. doi: 10.1034/j.1399-3038.2003.02085.x. PMID 12603707